CLINICAL TRIAL: NCT03778307
Title: Key Dimensions of Post-traumatic Stress Disorder (PTSD) and Endothelial Dysfunction (ED)
Brief Title: Key Dimensions of PTSD and ED
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jennifer A. Sumner, PhD, Assistant Professor, University of California, Los Angeles
Other Study IDs: AAAR8563; R01HL139614 (NIH)
Record Dates: First submitted 2018-12-07; First posted 2018-12-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Trauma; PTSD; Endothelial Dysfunction
Keywords: Trauma; PTSD; Endothelial Dysfunction
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and urine samples for inflammatory and oxidative stress biomarkers; a blood sample for DNA collection is an optional aspect of this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trauma exposed without PTSD: Individuals with a history of trauma exposure who do not have current PTSD
  Interventions: Behavioral: Psychophysiological fear conditioning and extinction task; Behavioral: Eyetracking task
- Trauma exposed with PTSD: Individuals with a history of trauma exposure and a current diagnosis of PTSD
  Interventions: Behavioral: Psychophysiological fear conditioning and extinction task; Behavioral: Eyetracking task

INTERVENTIONS:
Behavioral: Psychophysiological fear conditioning and extinction task — Behavioral task to assess psychophysiological measures of fear
Behavioral: Eyetracking task — Behavioral task to assess dysphoria-relevant attention allocation

SUMMARY:
This study will test whether endothelial dysfunction could be the early subclinical mechanism by which posttraumatic stress disorder (PTSD) increases cardiovascular disease (CVD) risk, and whether posttraumatic fear-a key component of PTSD-or another PTSD dimension could be the target to offset that risk. The results of this study may help trauma-exposed individuals who are at risk of having CVD events.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) increases risk of incident cardiovascular disease (CVD) by 25-50%. Most individuals (50-90%) experience a traumatic event in their lifetime, and PTSD is the fifth most common psychiatric disorder. Experts have now called for increased CVD surveillance after trauma and for PTSD treatment trials powered to reduce CVD risk. However, both CVD risk and PTSD are complex phenomena that likely interact in nuanced ways. This study will determine which PTSD dimension(s) contribute to endothelial dysfunction, one of the earliest modifiable precursors to CVD. The investigators will examine cross-sectional and longitudinal associations of PTSD and its underlying dimensions with functional and, secondarily, cellular measures of endothelial dysfunction (FMD and circulating endothelial cell-derived microparticles, respectively) in a community-dwelling sample of CVD-free adult men and women with a history of trauma (50% with current PTSD).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+ years
* History of exposure to a psychological trauma (e.g., natural disaster, physical assault)
* Fluent in English
* Willing to and capable of providing informed consent

Additional Inclusion Criteria for the PTSD Group

* Diagnosed with current PTSD (duration of at least 1 month) using the Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual 5th Edition (DSM-5) (CAPS-5) at the diagnostic interview assessment

Exclusion Criteria:

* History of CVD (i.e., diagnosis of myocardial infarction, unstable angina, heart failure, peripheral artery disease, or stroke)
* Deemed unable to comply with the protocol (either self-selected or by indicating during screening that could not complete all requested tasks)
* Current bipolar disorder or psychotic disorder
* Mild or more severe cognitive impairment [Mini-Mental State Exam (MMSE)3 score ≤18]
* Current moderate or severe substance use disorder
* Acute, unstable, or severe medical disorder or pregnancy
* Deemed to need immediate psychiatric intervention (e.g., active suicidality)
* Use of antipsychotic, mood stabilizer, antidepressant, or stimulant medication in the past 4 weeks
* Daily benzodiazepine use in the past 2 weeks

Additional Exclusion Criteria for the Trauma-Exposed Matched Control Group

* Current or past diagnosis of any DSM-5 psychiatric disorder
* CAPS-5 total score ≥25

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma-exposed adults without a history of cardiovascular disease recruited from the community
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation of the brachial artery (FMD) % | Baseline
  FMD is the percent difference in diameter of the brachial artery, before and after occlusion. Impaired endothelial function occurs when blood vessels are unable to dilate fully in response to nitric oxide synthesis and release, which is manifested as impaired endothelium-dependent vasodilation (i.e., lower FMD). Lower FMD has been associated with the degree of coronary atherosclerosis and predicts CVD events.

SECONDARY OUTCOMES:
Circulating EMPs expressing CD62E | Baseline
  EMPs expressing CD62E (i.e., endothelial cell activation) and CD31 (i.e., endothelial cell apoptosis) will be measured. Assessments of circulating EMPs will be measured using flow cytometry, and total flow cytometry counts will be converted to the number of EMPs per uL of blood. Higher concentrations of EMPs expressing CD62E and CD31 indicate greater endothelial dysfunction.
Circulating EMPs expressing CD31 | Baseline
  EMPs expressing CD62E (i.e., endothelial cell activation) and CD31 (i.e., endothelial cell apoptosis) will be measured. Assessments of circulating EMPs will be measured using flow cytometry, and total flow cytometry counts will be converted to the number of EMPs per uL of blood. Higher concentrations of EMPs expressing CD62E and CD31 indicate greater endothelial dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Sumner, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cleveland S, Reed K, Thomas JL, Ajijola OA, Ebrahimi R, Hsiai T, Lazarov A, Montoya AK, Neria Y, Shimbo D, Wolitzky-Taylor K, Sumner JA. Key dimensions of post-traumatic stress disorder and endothelial dysfunction: a protocol for a mechanism-focused cohort study. BMJ Open. 2021 May 5;11(5):e043060. doi: 10.1136/bmjopen-2020-043060. PMID 33952541